CLINICAL TRIAL: NCT05256628
Title: Early Versus Delayed Weightbearing in FemoroAcetabular Impingement Syndrome Patients Undergoing Treatment With Arthroscopic HIP Osteochondroplasty: a Randomized Controlled Non-inferiority Trial
Brief Title: Early Versus Delayed Weightbearing in Femoroacetabular Impingement Syndrome Patients
Acronym: FASTHIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Women's College Hospital (Other)
Collaborators: University of Toronto Orthopaedic Sports Medicine (Other)
Responsible Party: Principal Investigator, Dr. Tim Dwyer, Dr. Tim Dwyer, Orthopaedic Surgeon, Principal Investigator, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020-0154-B
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Femoroacetabular Impingement Syndrome
Keywords: Femoroacetabular Impingement; Femoroacetabular Impingement Syndrome; FAI; Hip Arthroscopy; Osteochondroplasty; Orthopaedics; Sports Medicine; Hip; Weight Bearing; Surgery; Arthroscopy
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Neither the patient nor their surgeon will be blinded. However, outcome assessors will be blinded throughout the duration of the study. Assessors will screen for complications at follow-up visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Weightbearing (Other): Patients randomized to early weightbearing will be permitted to begin immediate postoperative weightbearing as tolerated with crutches for additional stability.
  Interventions: Other: Early Weightbearing
- Protected Weightbearing (Other): Patients in the protected weightbearing group will be instructed to be touch weightbearing for a period of 6-weeks postoperatively before commencing to be weightbearing as tolerated.
  Interventions: Other: Protected Weightbearing

INTERVENTIONS:
Other: Early Weightbearing — Patients randomized to undergo this study intervention will bear weight, as tolerated, on the affected side straight after surgery, with crutches for additional support and stability. They will be allowed to stop using crutches in the weeks after surgery as they feel more comfortable and stable on their surgical leg.
  Arms: Early Weightbearing
Other: Protected Weightbearing — Patients randomized to undergo this study intervention will be instructed to be touch weightbearing for 6 weeks after surgery. They will use crutches and put no more weight on the surgical side than what it takes to crack an egg. After the 6-week mark, they will be able to bear weight.
  Arms: Protected Weightbearing

SUMMARY:
Femoroacetabular impingement syndrome (FAIS) is a condition caused by an abnormal bone structure that causes the bones on either side of the hip joint to impinge on each other during certain movements, thus causing pain. This condition can be surgically treated with hip arthroscopy. For patients undergoing hip arthroscopy, there are currently two protocols related to how they may bear their weight after surgery: 1) Delayed Weightbearing: Patients use crutches and put very little weight on the surgical side. After 6 weeks, they are able to bear weight, 2) Immediate Weightbearing: Patients bear weight on the affected side, as tolerated, immediately after surgery with crutches for additional support. They are then permitted to stop using the crutches in the weeks after surgery as they feel comfortable and are stable on the operative leg.

The purpose of this study is to determine whether immediate or delayed weightbearing protocols following hip arthroscopy impact patient outcomes and complication rates. Participants will be randomly allocated into one of the two aforementioned groups, and followed up for 2 years to assess function and patient-reported outcomes.

DETAILED DESCRIPTION:
Hip arthroscopy is used in the surgical treatment of femoroacetabular impingement syndrome (FAIS). There remains debate as to whether patients should be restricted to touch weightbearing post-operatively to prevent complications and improve clinical outcomes. This study aims to assess whether early weightbearing will produce non-inferior patient reported outcomes compared to protected touch weightbearing at 1 year post-operatively. We hypothesize that patients who are allowed to bear weight immediately after surgery will have non-inferior outcomes in comparison to those allowed to bear weight at 6 weeks post-operatively.

The FASTHIP trial is a multi-center, non-inferiority randomized controlled trial, looking at patients who are 16-50 years old, undergoing hip arthroscopy and osteochondroplasty for femoroacetabular impingement syndrome. All patients will be under general anesthesia, supine on a traction table. They will then undergo hip arthroscopy and associated procedures according to their respective surgeon's typical practice. This will result in different surgical techniques being represented in this study, with variances in portal placement, bone resection strategy, labral repair strategy and capsular closure technique. This is meant to reflect the true practice variances among hip arthroscopists and is inherent in the pragmatic nature of the trial. Participants will be randomized into one of two groups (immediate weightbearing as tolerated vs. touch weightbearing for 6 weeks following hip arthroscopy) in a 1:1 fashion using a computer-generated randomization schedule. Following surgery, all participants will receive a post-operative prescription of acetaminophen for three days, followed by Celebrex daily, and a conservative number of opioids for pain control. All participants will also receive standardized physiotherapy instructions outlining a phased approach from early joint protection and range of motion, to strengthening and sport specific goals in subsequent months. Initially, patients will be restricted to: hip extension 0, flexion 90, abduction 0, adduction 30 and limited external, internal rotation. At 6 weeks patients progress to full ROM and strengthening exercises. Return to sport targets instructions will be patient and sport specific, but generally recommended at 6 months.

Following screening, consent, collection of baseline data, and surgery, patients will be seen post-operatively at 2-weeks, 6-weeks, 3-months, 6-months, 1-year, and 2-years. Patient reported outcomes will be collected at 6 weeks, 3 months, 6-months, 1-year and 2-year appointments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of femoroacetabular impingement syndrome (FAIS)
* Booked for hip arthroscopy surgery and osteochondroplasty for FAIS at a participating site
* English literate

Exclusion Criteria:

* Prior hip surgery, arthroscopic or otherwise
* Workplace Safety and Insurance Board/medicolegal claim, complex regional pain syndrome, fibromyalgia, pain syndrome diagnoses, regular opioid use beyond 50mg morphine equivalents per day
* Hip dysplasia, Legg-Calve-Perthes disease or slipped capital femoral epiphysis, Arthritis > Tonnis 1
* Chondral matrix repair, microfracture/osteoarticular transfer system (OATS)

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
International Hip Outcome Tool (iHOT-33) | Administered at baseline, 6 months, 1 year, and 2 years post-operatively
  The primary outcome is the difference between the two interventions in their iHOT-33 scores at 1 year post-surgery.
  The iHOT-33 questionnaire consists of 33 questions evaluating hip symptoms, functional impairments, sporting activities, job concerns, as well as social and emotional wellbeing. Participants will rate their pain and impairment levels on a scale of 0 to 10, 0 being severe pain/impairment, and 10 being no pain or trouble at all.

SECONDARY OUTCOMES:
Hip Outcome Score, Activities of Daily Living (HOS-ADL) | Administered at baseline, 6 months, 1 year, and 2 years post-operatively
  The HOS-ADL consists of 17 questions that assess the impact of hip conditions on activities of daily living. Patients are asked to rate the level of difficulty in performing 17 different tasks, on a scale of 0 (unable to perform) to 4 (no difficulty at all).
European Quality of Life Five Dimension Five Level (EQ-5D-5L) | Administered at baseline, 6 months, 1 year, and 2 years post-operatively
  The EQ-5D-5L assesses patients' overall quality of life and health. This measure asks questions related to mobility, self-care, activity, pain, and anxiety/depression. The measure also includes one 0-100 scale assessing how patients perceive their overall health.
Pain Visual Analog Scale (VAS) | Administered at baseline, 2 weeks, 6 weeks, 3 months, 6 months, 1 year, and 2 years post-operatively
  Participants will indicate their level of pain on a 10cm line that represents a spectrum ranging from no pain (left side), to severe pain (right side)
Post-Operative Complications | Recorded at 2 weeks, 6 weeks, 3 months, 6 months, 1 year, and 2 years post-operatively.
  Incidences of complications such as infection, deep vein thrombosis, restrictions in ROM, adhesive capsulitis, fractures, prolonged opioid use, and early reoperation will be collected and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Dwyer, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colvin AC, Harrast J, Harner C. Trends in hip arthroscopy. J Bone Joint Surg Am. 2012 Feb 15;94(4):e23. doi: 10.2106/JBJS.J.01886. PMID 22336982
- [Background] Bozic KJ, Chan V, Valone FH 3rd, Feeley BT, Vail TP. Trends in hip arthroscopy utilization in the United States. J Arthroplasty. 2013 Sep;28(8 Suppl):140-3. doi: 10.1016/j.arth.2013.02.039. Epub 2013 Aug 1. PMID 23916639
- [Background] Montgomery SR, Ngo SS, Hobson T, Nguyen S, Alluri R, Wang JC, Hame SL. Trends and demographics in hip arthroscopy in the United States. Arthroscopy. 2013 Apr;29(4):661-5. doi: 10.1016/j.arthro.2012.11.005. Epub 2013 Feb 1. PMID 23375668
- [Background] Ross JR, Larson CM, Bedi A. Indications for Hip Arthroscopy. Sports Health. 2017 Sep/Oct;9(5):402-413. doi: 10.1177/1941738117712675. Epub 2017 Jul 5. PMID 28678628
- [Background] Ricciardi BF, Fabricant PD, Fields KG, Poultsides L, Zaltz I, Sink EL. What are the demographic and radiographic characteristics of patients with symptomatic extraarticular femoroacetabular impingement? Clin Orthop Relat Res. 2015 Apr;473(4):1299-308. doi: 10.1007/s11999-014-4001-3. PMID 25344401
- [Background] Petrera M, Yanez-Siller F, Whelan D, Hoit G, Mahjoob M, Chahal J, Dwyer T. Analysis of the referral pattern and wait time for hip arthroscopy in a single payer publicly funded health care system. J Eval Clin Pract. 2020 Feb;26(1):81-85. doi: 10.1111/jep.13192. Epub 2019 May 29. PMID 31144433
- [Background] Wylie JD, Peters CL, Aoki SK. Natural History of Structural Hip Abnormalities and the Potential for Hip Preservation. J Am Acad Orthop Surg. 2018 Aug 1;26(15):515-525. doi: 10.5435/JAAOS-D-16-00532. PMID 29939866
- [Background] McCarthy JC, Lee JA. History of hip arthroscopy: challenges and opportunities. Clin Sports Med. 2011 Apr;30(2):217-24. doi: 10.1016/j.csm.2010.12.001. PMID 21419953
- [Background] Collins JA, Ward JP, Youm T. Is prophylactic surgery for femoroacetabular impingement indicated? A systematic review. Am J Sports Med. 2014 Dec;42(12):3009-15. doi: 10.1177/0363546513499227. Epub 2013 Aug 21. PMID 23966568
- [Background] Ganz R, Parvizi J, Beck M, Leunig M, Notzli H, Siebenrock KA. Femoroacetabular impingement: a cause for osteoarthritis of the hip. Clin Orthop Relat Res. 2003 Dec;(417):112-20. doi: 10.1097/01.blo.0000096804.78689.c2. PMID 14646708
- [Background] Agricola R, Heijboer MP, Bierma-Zeinstra SM, Verhaar JA, Weinans H, Waarsing JH. Cam impingement causes osteoarthritis of the hip: a nationwide prospective cohort study (CHECK). Ann Rheum Dis. 2013 Jun;72(6):918-23. doi: 10.1136/annrheumdis-2012-201643. Epub 2012 Jun 23. PMID 22730371
- [Background] Cvetanovich GL, Lizzio V, Meta F, Chan D, Zaltz I, Nho SJ, Makhni EC. Variability and Comprehensiveness of North American Online Available Physical Therapy Protocols Following Hip Arthroscopy for Femoroacetabular Impingement and Labral Repair. Arthroscopy. 2017 Nov;33(11):1998-2005. doi: 10.1016/j.arthro.2017.06.045. Epub 2017 Sep 29. PMID 28969949
- [Background] Avnieli IB, Vidra M, Factor S, Atzmon R, Persitz J, Safran N, Rath E, Amar E. Postoperative Weightbearing Protocols After Arthroscopic Surgery for Femoroacetabular Impingement Does Not Affect Patient Outcome: A Comparative Study With Minimum 2-Year Follow-up. Arthroscopy. 2020 Jan;36(1):159-164. doi: 10.1016/j.arthro.2019.08.012. PMID 31864571
- [Background] Ayeni OR, Bedi A, Lorich DG, Kelly BT. Femoral neck fracture after arthroscopic management of femoroacetabular impingement: a case report. J Bone Joint Surg Am. 2011 May 4;93(9):e47. doi: 10.2106/JBJS.J.00792. No abstract available. PMID 21543668
- [Background] Weber AE, Harris JD, Nho SJ. Complications in Hip Arthroscopy: A Systematic Review and Strategies for Prevention. Sports Med Arthrosc Rev. 2015 Dec;23(4):187-93. doi: 10.1097/JSA.0000000000000084. PMID 26524553
- [Background] Mardones RM, Gonzalez C, Chen Q, Zobitz M, Kaufman KR, Trousdale RT. Surgical treatment of femoroacetabular impingement: evaluation of the effect of the size of the resection. J Bone Joint Surg Am. 2005 Feb;87(2):273-9. doi: 10.2106/JBJS.D.01793. PMID 15687147
- [Background] Alonso-Rasgado T, Jimenez-Cruz D, Bailey CG, Mandal P, Board T. Changes in the stress in the femoral head neck junction after osteochondroplasty for hip impingement: a finite element study. J Orthop Res. 2012 Dec;30(12):1999-2006. doi: 10.1002/jor.22164. Epub 2012 Jun 15. PMID 22707347
- [Background] Suchak AA, Bostick GP, Beaupre LA, Durand DC, Jomha NM. The influence of early weight-bearing compared with non-weight-bearing after surgical repair of the Achilles tendon. J Bone Joint Surg Am. 2008 Sep;90(9):1876-83. doi: 10.2106/JBJS.G.01242. PMID 18762647
- [Background] Tyler TF, McHugh MP, Gleim GW, Nicholas SJ. The effect of immediate weightbearing after anterior cruciate ligament reconstruction. Clin Orthop Relat Res. 1998 Dec;(357):141-8. doi: 10.1097/00003086-199812000-00019. PMID 9917711
- [Background] Smeeing DPJ, Houwert RM, Briet JP, Groenwold RHH, Lansink KWW, Leenen LPH, van der Zwaal P, Hoogendoorn JM, van Heijl M, Verleisdonk EJ, Segers MJM, Hietbrink F. Weight-bearing or non-weight-bearing after surgical treatment of ankle fractures: a multicenter randomized controlled trial. Eur J Trauma Emerg Surg. 2020 Feb;46(1):121-130. doi: 10.1007/s00068-018-1016-6. Epub 2018 Sep 24. PMID 30251154
- [Background] Andersson L, Wesslau A, Boden H, Dalen N. Immediate or late weight bearing after uncemented total hip arthroplasty: a study of functional recovery. J Arthroplasty. 2001 Dec;16(8):1063-5. doi: 10.1054/arth.2001.27253. PMID 11740764
- [Background] Rath E, Sharfman ZT, Paret M, Amar E, Drexler M, Bonin N. Hip arthroscopy protocol: expert opinions on post-operative weight bearing and return to sports guidelines. J Hip Preserv Surg. 2017 Feb 23;4(1):60-66. doi: 10.1093/jhps/hnw045. eCollection 2017 Jan. PMID 28630722
- [Background] Koh JL, Gupta K. Evaluation of repair of the hip labrum under simulated full weight-bearing. Hip Int. 2017 Feb 21;27(1):104-109. doi: 10.5301/hipint.5000472. Epub 2017 Jan 24. PMID 28127741
- [Background] Griffin DR, Dickenson EJ, O'Donnell J, Agricola R, Awan T, Beck M, Clohisy JC, Dijkstra HP, Falvey E, Gimpel M, Hinman RS, Holmich P, Kassarjian A, Martin HD, Martin R, Mather RC, Philippon MJ, Reiman MP, Takla A, Thorborg K, Walker S, Weir A, Bennell KL. The Warwick Agreement on femoroacetabular impingement syndrome (FAI syndrome): an international consensus statement. Br J Sports Med. 2016 Oct;50(19):1169-76. doi: 10.1136/bjsports-2016-096743. PMID 27629403
- [Background] Gwathmey FW, Jones KS, Thomas Byrd JW. Revision hip arthroscopy: findings and outcomes. J Hip Preserv Surg. 2017 May 11;4(4):318-323. doi: 10.1093/jhps/hnx014. eCollection 2017 Dec. PMID 29250340
- [Background] Palmer S, Bailey J, Brown C, Jones A, McCabe CS. Sensory Function and Pain Experience in Arthritis, Complex Regional Pain Syndrome, Fibromyalgia Syndrome, and Pain-Free Volunteers: A Cross-Sectional Study. Clin J Pain. 2019 Nov;35(11):894-900. doi: 10.1097/AJP.0000000000000751. PMID 31408010
- [Background] Murgatroyd DF, Casey PP, Cameron ID, Harris IA. The effect of financial compensation on health outcomes following musculoskeletal injury: systematic review. PLoS One. 2015 Feb 13;10(2):e0117597. doi: 10.1371/journal.pone.0117597. eCollection 2015. PMID 25680118
- [Background] Nabavi A, Olwill CM, Harris IA. Preoperative predictors of outcome in the arthroscopic treatment of femoroacetabular impingement. Hip Int. 2015 Sep-Oct;25(5):402-5. doi: 10.5301/hipint.5000261. Epub 2015 May 27. PMID 26044534
- [Background] Kemp JL, MacDonald D, Collins NJ, Hatton AL, Crossley KM. Hip arthroscopy in the setting of hip osteoarthritis: systematic review of outcomes and progression to hip arthroplasty. Clin Orthop Relat Res. 2015 Mar;473(3):1055-73. doi: 10.1007/s11999-014-3943-9. Epub 2014 Sep 18. PMID 25231154
- [Background] Philippon MJ, Briggs KK, Carlisle JC, Patterson DC. Joint space predicts THA after hip arthroscopy in patients 50 years and older. Clin Orthop Relat Res. 2013 Aug;471(8):2492-6. doi: 10.1007/s11999-012-2779-4. PMID 23292888
- [Background] Mohtadi NG, Griffin DR, Pedersen ME, Chan D, Safran MR, Parsons N, Sekiya JK, Kelly BT, Werle JR, Leunig M, McCarthy JC, Martin HD, Byrd JW, Philippon MJ, Martin RL, Guanche CA, Clohisy JC, Sampson TG, Kocher MS, Larson CM; Multicenter Arthroscopy of the Hip Outcomes Research Network. The Development and validation of a self-administered quality-of-life outcome measure for young, active patients with symptomatic hip disease: the International Hip Outcome Tool (iHOT-33). Arthroscopy. 2012 May;28(5):595-605; quiz 606-10.e1. doi: 10.1016/j.arthro.2012.03.013. PMID 22542433
- [Background] Griffin DR, Parsons N, Mohtadi NG, Safran MR; Multicenter Arthroscopy of the Hip Outcomes Research Network. A short version of the International Hip Outcome Tool (iHOT-12) for use in routine clinical practice. Arthroscopy. 2012 May;28(5):611-6; quiz 616-8. doi: 10.1016/j.arthro.2012.02.027. PMID 22542434
- [Background] Kemp JL, Collins NJ, Roos EM, Crossley KM. Psychometric properties of patient-reported outcome measures for hip arthroscopic surgery. Am J Sports Med. 2013 Sep;41(9):2065-73. doi: 10.1177/0363546513494173. Epub 2013 Jul 8. PMID 23835268
- [Background] Griffin D, Wall P, Realpe A, Adams A, Parsons N, Hobson R, Achten J, Fry J, Costa M, Petrou S, Foster N, Donovan J. UK FASHIoN: feasibility study of a randomised controlled trial of arthroscopic surgery for hip impingement compared with best conservative care. Health Technol Assess. 2016 Apr;20(32):1-172. doi: 10.3310/hta20320. PMID 27117505
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Devlin NJ, Shah KK, Feng Y, Mulhern B, van Hout B. Valuing health-related quality of life: An EQ-5D-5L value set for England. Health Econ. 2018 Jan;27(1):7-22. doi: 10.1002/hec.3564. Epub 2017 Aug 22. PMID 28833869
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Cvetanovich GL, Chalmers PN, Levy DM, Mather RC 3rd, Harris JD, Bush-Joseph CA, Nho SJ. Hip Arthroscopy Surgical Volume Trends and 30-Day Postoperative Complications. Arthroscopy. 2016 Jul;32(7):1286-92. doi: 10.1016/j.arthro.2016.01.042. Epub 2016 Apr 9. PMID 27067059
- [Background] Nakano N, Khanduja V. Complications in Hip Arthroscopy. Muscles Ligaments Tendons J. 2016 Dec 21;6(3):402-409. doi: 10.11138/mltj/2016.6.3.402. eCollection 2016 Jul-Sep. PMID 28066747
- [Background] Julious SA. Sample sizes for clinical trials with normal data. Stat Med. 2004 Jun 30;23(12):1921-86. doi: 10.1002/sim.1783. PMID 15195324